CLINICAL TRIAL: NCT06549348
Title: Radiation Free Study
Acronym: RadFree
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IGT-00915-RadFree
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Task navigation using fluoroscopy guidance (No Intervention): Standard of care treatment using
- Task navigation using LumiGuide (Active Comparator): Standard of care treatment using LumiGuide fluoroscopy guidance
  Interventions: Radiation: Measure average procedure fluoroscopy time using LumiGuide and conventional fluoroscopy guidance

INTERVENTIONS:
Radiation: Measure average procedure fluoroscopy time using LumiGuide and conventional fluoroscopy guidance — Fenestrated Endovascular Aortic Repair (FEVAR) procedure done with either LumiGuide or conventional fluoroscopy guidance
  Arms: Task navigation using LumiGuide

SUMMARY:
This is a prospective, randomized, unblinded, multi-center study. Sites were selected from different geographies (EU and US) with different clinical practice to ensure the results are more generalizable.

Primary objective is to demonstrate that the average procedure fluoroscopy time using LumiGuide is lower compared to conventional fluoroscopy guidance in Fenestrated Endovascular Aortic Repair (FEVAR)

ELIGIBILITY:
Inclusion Criteria:

* Subject will be undergoing a primary Fenestrated Endovascular Aortic Repair (FEVAR) procedure (including subjects with prior infrarenal EVAR or open repair) that includes the incorporation of visceral arteries into the repair.
* Subject is able to give informed consent and is 18 years of age or older, or of legal age to give informed consent per state or national law.
* Subject has a life expectancy of at least 2 years
* Target vessels to be included are the Celiac Trunk, Superior Mesenteric Artery and Renal Arteries

Exclusion Criteria:

* Subjects undergoing an endovascular procedure that include branches or iliac branched devices (IBD) in the repair
* Subject treated for re-intervention / staged procedure post-primary FEVAR procedure
* Subjects intended to be treated for more than 4 target vessels (not counting the contralateral gate)
* Subject treated for an emergent (<24hrs after emergence) procedure
* Subject with connective tissue disorder eg, Marfan's or Ehlers Danlos Syndrome
* Subject with contrast allergies
* Subject participates in a potentially confounding drug or device trial during the course of the study. Co-enrollment in concurrent trials may be allowed provided that pre-approval is obtained from Philips.
* All vulnerable subjects such as immuno-compromised subjects, subjects lacking the capacity to provide consent, patients in emergency situations, pregnant or breast-feeding women, or any other subject who meets an exclusion criteria, according to applicable national laws, if any.
* Subject unwilling or unable to comply with the protocol unable to understand verbal and/or written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that the average procedure fluoroscopy time using LumiGuide is lower compared to conventional fluoroscopy guidance in Fenestrated Endovascular Aortic Repair (FEVAR). | Fenestrated Endovascular Aortic Repair (FEVAR) procedure (skin to skin procedure time)
  Procedure fluoroscopy time

CONTACTS AND LOCATIONS:
Locations (9):
- United States (4):
  - University of Alabama, Birmingham, Alabama
  - University of Massachusetts, Worcester, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
- UZ Gent, Ghent, Belgium
- Rigshospitalet University Hospital, Copenhagen, Denmark
- Hôpital Universitaire Pitié-Salpêtrière, Paris, France
- UMC Maastricht, Maastricht, Netherlands
- Guys & St Thomas, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No